CLINICAL TRIAL: NCT01084811
Title: Chronic Rhinosinusitis: Biochemical Markers and Biofilm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Erik S Lie, University Hospital, Akershus
Other Study IDs: 2009/1720(REK)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Rhinosinusitis
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal mucosa and nasal polyps
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chronic rhinosinusitis with nasal polyps
  Interventions: Procedure: biopsy
- chronic rhinosinusitis without nasal polyps
  Interventions: Procedure: biopsy
- Control group
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — One or more biopsies from nasal mucosa will be harvested during surgery

SUMMARY:
The investigators will conduct a descriptive, prospective, three-armed study concerning the pathophysiology of chronic rhinosinusitis.

In one part of the study the investigators want to investigate the presence of biofilm in patients with chronic rhinosinusitis both with and without nasal polyps compared with a control group of subjects without chronic rhinosinusitis. The investigators will also compare quality of life in the three groups and correlate disease severity in biofilm patients versus patients where biofilm was not present.

The hypothesis here is that biofilm patients suffers a more severe disease.

In the other arm of the study the investigators will compare the presence of different biochemical compounds in the three study groups. The investigators specifically want to investigate matrix metalloproteases and apoptosis-inhibitors with immunohistochemistry. The investigators may also add other compounds to our test-battery if interesting candidates surface in the literature during the inclusion period.

The purpose of this part of the study is to investigate candidates for the development of nasal polyposis.

The investigators plan to include 100 patients suffering from chronic rhinosinusitis with nasal polyps, and 100 patients with chronic rhinosinusitis without nasal polyps and 30 control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis based on EPOS3
* Submitted to surgery
* Using nasal corticosteroids

Exclusion Criteria:

* Age below 18 years
* Using antibiotics at the time of surgery
* Using systemic corticosteroids
* Sempers triad

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to sinonasal surgery at Ahus, Norway
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahus, Lørenskog, Akershus, Norway